CLINICAL TRIAL: NCT03074578
Title: Y a T-il Une désensibilisation Pendant le Sommeil après la réception de Violence Verbale ?
Brief Title: Is There a Desensitization During Sleep After Exposure to a Violent Verbal Input ?
Acronym: COREV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre National de la Recherche Scientifique, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Isabelle Arnulf, Professor, Centre National de la Recherche Scientifique, France
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 16009; COREV (Other: Centre d'Investigation Clinique Paris-Est)
Record Dates: First submitted 2017-03-01; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Verbal Abuse
Keywords: sleep; verbal abuse; polysomnography; perception; neuropsychological tests

STUDY DESIGN:
Intervention Model Description: Watching two different videos (one violent, one non-violent), re-exposure after 11h daytime (wake period) or 11h nighttime (sleep period). The order of videos is balanced, in a cross over fashion
Who Masked: Outcomes Assessor
Masking Description: The analysis of heart signal, polysomnography and dream reports analysis will be performed by assessors masked to the group and type of video.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Night-time desensitization (Experimental): Watching a video containing verbal and visual violence in the evening, and again in the next morning
  Interventions: Behavioral: Watching Video-clip 1; Behavioral: Watching Video-clip 2
- Daytime desensitization (Sham Comparator): Watching a video containing verbal and visual non-violence in the morning, and then again the evening of the same day
  Interventions: Behavioral: Watching Video-clip 1; Behavioral: Watching Video-clip 2

INTERVENTIONS:
Behavioral: Watching Video-clip 1 — Video -clip 1 contains violent images and text
Behavioral: Watching Video-clip 2 — Video -clip 2 contains neutral images and text

SUMMARY:
There is a need for quantify the emotional and neurophysiological perception of verbal violence, in order to understand the impact it might have on a subject. This project aims at assessing the influence of time, sleep, and people interaction on the perception of verbal violence.

DETAILED DESCRIPTION:
There are many processes involved in the perception of verbal violence. There is a need for quantified data to have a better understanding the physiological and neurological perception of verbal violence, in order to understand the impact it might have on a subject. This project aims at assessing the influence of time, sleep, and people interaction on the perception of verbal violence. The "cognitive replay" will also be assessed through dreams. The investigators think that sleep plays a role in desensitization to negative emotions and to memory consolidation. However, the role of sleep in verbal violence remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Subject fully understands French
* Subject willing to consent to the study and signed the written consent
* Subject is afiliated to the Freanch national health care system (Sécurité Sociale)
* Subject level of education superior to "Brevet des collèges" (an equivalent would be the general certificate of secondary education)

Exclusion Criteria:

* The subject is not able to understand the protocol
* The subject has a language disorder
* The subject has a psychiatric or neurological disorders
* The subject does not use psychotropic drugs
* The subject has watched the advertidement : "stop djihadisme", broadcasted on television by the french government

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate | During each video exposure (duration 1.2 min), 4 times
  heart rate in beat per min

SECONDARY OUTCOMES:
Sweating | During the video exposure (duration 1.2 min), 4 times
  measure of electrodermal reaction, in millivolts
Vasoconstriction | During the video exposure (duration 1.2 min), 4 times
  measure of the pulse wave, in millivolts
Emotions | Just after the video exposure, during 1 min
  Analogic visual scales, in mm

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnulf, MD, PhD, Principal Investigator — Pitie Salpêtrière Hospital, Paris, France
Locations (1):
- Service des pathologies du sommeil, Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barros A, Uguccioni G, Salkin-Goux V, Leu-Semenescu S, Dodet P, Arnulf I. Simple behavioral criteria for the diagnosis of disorders of arousal. J Clin Sleep Med. 2020 Jan 15;16(1):121-128. doi: 10.5664/jcsm.8136. Epub 2019 Dec 4. PMID 31957639